CLINICAL TRIAL: NCT04622397
Title: Local Subfascial and Intramuscular Tranexamic Acid Administration in Pediatric Patient Undergoing Scoliosis Surgery, Double Blind Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: tranexamic acid in scoliosis
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Blood Loss, Surgical; Scoliosis
MeSH Terms: conditions — Blood Loss, Surgical; Scoliosis | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: randomized comparative study
Who Masked: Care Provider
Masking Description: surgeon will be blinded to type of injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (tranexamic acid),n=15 (Active Comparator): Group T: tranexamic acid 10 mg/kg will be injected locally
  Interventions: Drug: Tranexamic acid injection
- Group S (saline) (n=15) (Placebo Comparator): Group S saline will be injected
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic acid injection — Local subfascial and intramuscular infiltration will be performed by surgeon at levels of fixation prior to skine incision
  Arms: Group T (tranexamic acid),n=15
Drug: Saline — Local subfascial and intramuscular infiltration will be performed by surgeon at levels of fixation prior to skine incision
  Arms: Group S (saline) (n=15)

SUMMARY:
We hypothesized that local administration of tranexamic acid will minimize blood loss and blood product administration in pediatric patient undergoing scoliosis surgery

DETAILED DESCRIPTION:
Spine surgery in paediatrics is frequently associated with substantial blood loss.

Blood product adminestration in children has many complications that are not fully known.

There are many modalities currently available to reduce blood loss in pediatric patients.

Tranexamic acid is tissue plasminogen activator inhibitor that reduce perioperative blood loss.

To date, no studies have investigated effect of local administration of tranexamic acid in pediatric population undergoing scoliosis surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-12 years
* Of both sexes
* American society of anesthesiologist (ASA) physical status classification class I
* Undergoing general anesthesia for scoliosis surgery

Exclusion Criteria:

* Parents' refusal of regional block
* Known allergy to tranexamic acid
* Bleeding disorders (INR >1.4,Platelet count< 75000)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2021-11-29 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Intraperative blood loss in both groups | period of surgery(1-2 hours)
  amount of blood/kg(ml/kg)

SECONDARY OUTCOMES:
post-operative blood loss | 24 hours
  amount of blood in drain after surgery
Blood product admenestration | duration of procedure(1-2 hours)
  units of blood given during surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bible JE, Mirza M, Knaub MA. Blood-loss Management in Spine Surgery. J Am Acad Orthop Surg. 2018 Jan 15;26(2):35-44. doi: 10.5435/JAAOS-D-16-00184. PMID 29303921
- [Background] Goobie SM. A blood transfusion can save a child's life or threaten it. Paediatr Anaesth. 2015 Dec;25(12):1182-3. doi: 10.1111/pan.12816. No abstract available. PMID 26507915
- [Background] Mikhail C, Pennington Z, Arnold PM, Brodke DS, Chapman JR, Chutkan N, Daubs MD, DeVine JG, Fehlings MG, Gelb DE, Ghobrial GM, Harrop JS, Hoelscher C, Jiang F, Knightly JJ, Kwon BK, Mroz TE, Nassr A, Riew KD, Sekhon LH, Smith JS, Traynelis VC, Wang JC, Weber MH, Wilson JR, Witiw CD, Sciubba DM, Cho SK. Minimizing Blood Loss in Spine Surgery. Global Spine J. 2020 Jan;10(1 Suppl):71S-83S. doi: 10.1177/2192568219868475. Epub 2020 Jan 6. PMID 31934525
- [Background] Slaughter TF, Greenberg CS. Antifibrinolytic drugs and perioperative hemostasis. Am J Hematol. 1997 Sep;56(1):32-6. doi: 10.1002/(sici)1096-8652(199709)56:13.0.co;2-3. PMID 9298865